CLINICAL TRIAL: NCT02423564
Title: A Double-blind, Placebo-controlled, Parallel Study Investigating the Effect of Digesta-Lac in Healthy Adults With Occasional Constipation
Brief Title: A Study Investigating the Effect of Digesta-Lac in Healthy Adults With Occasional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Global Institute of Probiotics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 14PCHN
Record Dates: First submitted 2015-04-13; First posted 2015-04-22 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Occasional Constipation
Keywords: Probiotic; Digesta-Lac; Occasional Constipation; Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Population with Digesta Lac (Active Comparator): Digesta Lac is Lactobacillus bulgaricus LB-51 at 2.0 billion cfu with non-medicinal ingredients: cellulose, potato powder, chick pea extract, vitamin c, L-leucine, vegetable capsule (hypromellose)
  Interventions: Dietary Supplement: Digesta Lac
- Healthy Population with Placebo (Placebo Comparator): Placebo contains: cellulose, Organic Whole Grain Brown Rice Milk Concentrate, L-Leucine, potato powder, vegetable capsule (hypromellose)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Digesta Lac
  Arms: Healthy Population with Digesta Lac
Other: Placebo
  Arms: Healthy Population with Placebo

SUMMARY:
This investigation will evaluate the effect of Digesta-Lac in adults with occasional constipation in a single-center, randomized, double-blind, placebo-controlled, parallel group 2-arm study for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18-65 years of age (inclusive)
* If female, subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

OR Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include: Double barrier method, Hormonal contraceptives (including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)), Intrauterine devices, Vasectomy of partner, Non-heterosexual lifestyle

* BMI 18.5-35.0kg/m2
* Subjects must have < 3 bowel movements per week for at least 2 weeks (but for not more than 12 weeks in the past 6 months) prior to randomization (confirmed at screening and baseline) and the presence of at least one other bowel symptom of constipation in at least 25% of defecations; Hard stools. or complete lack of loose or watery stools, straining during defecation, feelings of incomplete evacuation, abdominal discomfort, bloating/distension
* Healthy as determined by laboratory results, medical history and physical exam
* Subjects must agree not to use any other products or therapies (i.e. enemas) to treat their constipation during the run-in to the study (7 days prior to baseline) or during the course of the study except as a rescue medication.
* Agrees not to change current dietary habits (with the exception of avoiding pro- and prebiotics), smoking habits and activity/training levels one week prior to randomization and during the course of the study
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Subjects currently under a doctor's care and treatment for constipation
* Subjects that have a history of chronic constipation(defined as <3 bowel movements per week for more than 3 months) due to any underlying cause (IBS, functional constipation [chronic constipation], IBD, ulcer, etc.) based on self-report, physical examination, or documented medical history
* Subjects who have severe abdominal pain as the predominant constipation symptom as determined by the Principal Investigator.
* Subjects who have a history of colorectal cancer, anal abscess, anal fistula, anal fissure, anal stenosis, gastric retention or obstruction, bowel resection, rectocele, colostomy, IBS, Crohn's disease, episiotomy or hemorrhoids.
* Subjects with a history of spinal injuries and/or surgeries which could result in an atonic colon or saddle anesthesia (i.e. spinal fusion in the lumbar spine)
* Subjects who have been hospitalized within the past 3 months
* Subjects with known renal or hepatic insufficiency
* Subjects with gastrointestinal bleeding or acute infection
* Subjects who use prescription medication to treat constipation
* Subjects who have previously suffered from slipped discs
* Subjects who plan to use OTC laxatives or stool softeners, or any other products meant to treat constipation other than the study supplements, during the treatment period (use as a rescue medication is permitted) or other therapies such as enemas.
* Subjects currently taking or taken within 28 days of randomization a concomitant medication that causes constipation which in the Principle Investigator's opinion may impact the study results.
* Any non-gastrointestinal disease/complication that, in the investigator's opinion, may affect subject safety or confound the evaluation of the study endpoints
* Immunodeficiency (i.e. HIV positive, rheumatoid arthritis, history of organ transplant)
* Clinically significant abnormal laboratory results at screening (e.g. AST and/or ALT > 2 x ULN, and/or bilirubin > 2 x ULN; serum creatinine > 1.5 x ULN; hemoglobin < 140 g/L for males and < 123 g/L for females)
* Abdominal or perineal surgery within 6 months of randomization
* Subjects who plan on engaging in anal intercourse during the run-in or treatment periods of the trial. Enemas are not allowed within 7 days of randomization or throughout the trial.
* Participation in a clinical research trial within 30 days prior to randomization or participation in a clinical trial researching a probiotic within 60 days prior to randomization
* Currently taking anti-psychotic medication
* Allergy or sensitivity to study supplement ingredients
* Use of pre- and probiotics within 8 weeks prior to randomization
* Alcohol abuse (>2 standard alcoholic drinks per day) or drug abuse within the past 6 months
* Individuals who are cognitively impaired and/or who are unable to give informed consent.
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mean difference (probiotic - placebo) in the number of weekly complete spontaneous bowel movements | Baseline to Day 21

SECONDARY OUTCOMES:
The between group difference in the average number of weekly complete spontaneous bowel movements | Baseline to Day 21
The percentage of responders vs. non- responders for the average number of weekly complete spontaneous bowel movements | Day 21
The mean difference (probiotic - placebo) in the number of weekly spontaneous bowel movements | Baseline to Day 21
The between group difference in the average number of weekly spontaneous bowel movements | Baseline to Day 21
The percentage of responders vs. non- responders for the average number of weekly spontaneous bowel movements | Day 21
The mean difference (probiotic - placebo) in the number of weekly bowel movements | Baseline to Day 21
The between group difference in the average number of weekly bowel movements | Baseline to Day 21
The percentage of responders vs. non- responders for the average number of weekly bowel movements | Day 21
Changes in bowel habits (straining, feeling of complete evacuation) as assessed by the daily bowel habits diary | Baseline to Day 21
Change in Bristol Stool Score | Baseline to Day 21
Change in symptoms related to constipation determined by the Gastrointestinal Symptom Rating Scale | Baseline to Day 21
Mean score of the Product Perception Questionnaire | Day 21
The between group difference in the percentage of subjects that used a laxative | Baseline to Day 21
The between group difference in the total number of days per subject that a laxative | Baseline to Day 21

OTHER OUTCOMES:
Laboratory parameters of safety - CBC | Screening to Day 21
Laboratory parameters of safety - Electrolytes | Screening to Day 21
Laboratory parameters of safety - Kidney function markers | Screening to Day 21
Laboratory parameters of safety - Liver function markers | Screening to Day 21
Anthropometric measures - Weight | Screening to Day 21
Anthropometric measures - BMI | Screening to Day 21
Anthropometric measures - Blood Pressure | Screening to Day 21
Anthropometric measures - Heart Rate | Screening to Day 21
Incidence of Adverse Events | Baseline to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada